CLINICAL TRIAL: NCT02543320
Title: Neurofeedback for Acute Radiotherapy-Induced Pain in Head and Neck Cancer Patients
Brief Title: Neurofeedback in Decreasing Acute Radiotherapy-Induced Pain in Patients With Head and Neck Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-1102; NCI-2017-00521 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-1102 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (neurofeedback) (Experimental): Beginning at weeks 4 and 5 or 5 and 6 of radiotherapy, patients undergo neurofeedback training QID TIW for up to 6 treatments. Patients also complete questionnaires over 10 minutes at baseline and after neurofeedback training.
  Interventions: Other: LORETA Neurofeedback Training; Other: Questionnaire Administration

INTERVENTIONS:
Other: LORETA Neurofeedback Training — Undergo LORETA neurofeedback training
  Other Names: LNFB Training; LORETA Neurofeedback; LORETA Z-score Neurofeedback Training; LORETA Z-score NFT; LORETA Z-score Training; LORETA-EEG-NFB; Low Resolution Electromagnetic Tomography Neurofeedback Training; LZNFT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot trial studies how well neurofeedback training works in decreasing acute radiotherapy-induced pain in patients with head and neck cancer. Neurofeedback training is a type of therapy that uses electroencephalograph and a computer software program to measure brain wave activity. Neurofeedback training may help teach patients ways to modify their own brain waves to decrease the perception of pain and improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effects of an individualized LORETA (low resolution electromagnetic tomography) Z score neurofeedback program on changes in brain function using EEG (electroencephalography), qEEG (quantitative electroencephalography), and LORETA from immediately before to after each session in patients with head and neck cancer undergoing radiotherapy and experiencing pain.

SECONDARY OBJECTIVES:

I. Examine the effects of an individualized LORETA Z score neurofeedback program on perceptions of radiation-induced pain in head and neck cancer patients from immediately before neurofeedback training to immediately after neurofeedback training.

II. Identify brain regions from qEEG and LORETA that are associated with a non-pain state and then an acute pain state.

III. Examine the relationship between the patient and their spouse or primary caregiver.

OUTLINE:

Beginning at weeks 4 and 5 or 5 and 6 of radiotherapy, patients undergo neurofeedback training once per day (QID) three times per week (TIW) for up to 6 treatments. Patients also complete questionnaires over 10 minutes at baseline and after neurofeedback training.

After completion of study, patients are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and read English, sign a written informed consent, and be willing to follow protocol requirements
* Patients must not have pain > 2 on a scale of 0 - 10 (self report) in the head and neck before starting radiotherapy
* Scheduled to undergo a 6 week course of radiotherapy for head and neck cancer
* No plans to change the type of pain medication during the course of the study

Exclusion Criteria:

* Patients who are taking any antipsychotic medications
* Patients with active central nervous system (CNS) disease, such as clinically-evident metastases or leptomeningeal disease, dementia, or encephalopathy
* Patients who have ever been diagnosed with bipolar disorder or schizophrenia
* Patients with known, previously diagnosed head or neck pain from other pain syndromes or chronic pain requiring analgesics
* Patients with a history of seizure disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08-29 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
EEG | Baseline up to 1 week
  The qEEG normative database is grouped by age and contains a sufficiently large sample size with means and standard deviations of the EEG time series and/or frequency domain analysis computed for each age group.
Neurofeeback (LORETA) | Up to 5 years
  The LORETA software package is used to perform the statistical analyses. The methodology used is non-parametric. It is based on estimating, via randomization, the empirical probability distribution for the max-statistic (e.g. the maximum of a t or an F statistic), under the null hypothesis. This methodology corrects for multiple testing (i.e., for the collection of tests performed for all electrodes and/or voxels, and for all time samples and/or discrete frequencies. Due to the non-parametric nature of the method, its validity need not rely on any assumption of Gaussianity.

SECONDARY OUTCOMES:
The Brief Pain Inventory (Short Form) | Up to 5 years
  is a validated, widely used, self-administered questionnaire to assess severity of pain and impact of pain on daily functioning among patients (Cleeland, 2006; Cleeland, 1991; Tan, 2004). The Brief Pain Inventory (Short form) Scale 0-10 (No Pain 0-10 As Bad as you can imagine ).
The Multidimensional Pain Inventory (MPI) | Up to 5 years
  is a measure generally used in chronic pain conditions used to measure the patient perception of their pain experience. The MPI has 4 subscales that assess pain intensity, emotional distress, cognitive and functional adaptation, and social support. It is used to assess overall adjustment of pain and outcomes of treatment interventions. Although it is generally used for chronic pain patients, the MPI has also been used in studies with patients who have acute pain (Edwards, Et al., 2006; Montes Doncel, et al., 2001).
The Social Provisions Scale (SPS) | Up to 5 years
  will also be administered with the MPI as a measure of validity. The inclusion of these measures allows us to assess perceived relational support in general (SPS) and in specific relation to their pain (MPI). For the patients who consent to their spouses/caregivers participating in the optional survey, the spouses/caregivers will be given the SPS at the same timepoints as the patient.
M. D. Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN): | Up to 5 years
  Cancer-related symptoms will be assessed using the validated MDASI-HN. The MDASI measures, on a numeric rating scale of 0-10, both the severity of symptoms and the interference symptoms cause in patients" daily activities. The 13 core MDASI symptom items are based on extensive evaluation of symptoms common to cancer and cancer treatment. The MDASI-HN includes 9 head and neck-specific items. The instrument was validated in a cohort of more than 200 patients and found to be highly reliable (Rosenthal, Mendoza, & Chambers, 2007).
Visual analog scale to assess pain | Up to 5 years
  A visual analog scale to assess pain (0-10 scale) will be used before and after each training session to determine if change in brain function is meaningful clinically.
  A visual analog scale to assess mouth sores (0-10 scale) will be used before each training session to determine patient perception of interference with quality of life due to mucositis. A visual analog scale to assess patient comfort (0-10 scale) will be used before and after each training session to determine patient perception of overall comfort.
Pain medication use | Up to 5 years
  All medications prescribed and used by the patients for pain or other medical conditions will be collected during the time they are participating in the study. We will use descriptive statistics to summarize pain medication use over the course of the study and radiation dose. We will tabulate adverse events by grade and relationship to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Prinsloo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org